CLINICAL TRIAL: NCT03223220
Title: Quelling of Excitotoxicity in Acute Stroke With Ketamine
Acronym: QUEST-KETA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lower Merion Neurology Research Foundation (Other)
Responsible Party: Principal Investigator, Sudhir Aggarwal MD, PhD,, Neurologist and Medical Director, Lower Merion Neurology Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LMNRF-001
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke, Neuroprotection, Ketamine
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Ketamine; Saline Solution; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug (Experimental): Will receive Ketamine infusion, and Midazolam (Versed).
  Interventions: Drug: Ketamine; Drug: Midazolam injection
- Placebo (Placebo Comparator): Will receive Normal saline infusion and Midazolam (Versed).
  Interventions: Other: Normal Saline; Drug: Midazolam injection

INTERVENTIONS:
Drug: Ketamine — IV infusion
  Arms: Study Drug
Other: Normal Saline — IV infusion
  Arms: Placebo
Drug: Midazolam injection — Injection
  Other Names: Versed

SUMMARY:
The investigators plan to undertake a phase II study to investigate the efficacy and side effects of intravenous ketamine to reduce neuroexcitotoxicity, and thus provide neuroprotection in patients diagnosed with acute ischemic stroke.

DETAILED DESCRIPTION:
After obtaining informed consent, patients enrolled in the 'study drug' arm of the trial will receive Ketamine (1 mg/ml solution prepared in normal saline) infusion at a rate of 20 mg/h for a period of 24 hours. The infusion will start at a rate of 5 mg/h, and then gradually tapered up during the first 3 hours by 5 mg an hour. Similarly, the infusion rate will be gradually tapered down at a rate of 5 mg/h during the last 3 hours of infusion. The patients randomized to the 'placebo arm' of the trial will receive normal saline infusion at the same rates. In order to prevent the psychogenic adverse effects associated with Ketamine, the patients will be administered Midazolam at a dose of 1 mg IV every 4 hours. Midazolam will also be administered at the same rate to the patients randomized to the placebo arm. Blood Ketamine levels will be measured before starting the treatment, and daily while the infusion is on. While receiving treatment, the patients will be admitted to the telemetry floor in the hospital, on a monitored bed.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who are 18 years or older, presenting or admitted to the study site with acute ischemic stroke, up to 24 hours since their last known well time
2. An MRI evidence of acute ischemic infarct on the diffusion-weighted imaging with ADC correlate
3. Pre-stroke modified Rankin scale of 0-2
4. Patient should be willing to participate in the study by providing a written consent himself/herself or through a proxy.

Exclusion Criteria:

1. Eligibility to receive IV Alteplase or intra-arterial thrombectomy/embolectomy
2. Longer than 24 hours since last known well time
3. Pre-stroke modified Rankin scale of 3 or above.
4. Pregnant or lactating females
5. Pre-existing psychiatric illness
6. Intracranial hemorrhage of any type at presentation
7. Seizure at onset of symptoms
8. Sustained uncontrolled hypertension defined as Systolic Blood pressure greater than 185 mmHg or Diastolic Blood Pressure greater than 110 mmHg, despite administration of antihypertensive medications
9. Known hypersensitivity or adverse reaction to prior administration of Ketamine
10. Inability/refusal to provide consent by the patient or through a proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in weighted modified Rankin scale score between day 1 and 90 will be assessed. | On day 1 and at 90 days
  An improvement of 2 in mRS score will be considered favorable outcome.

SECONDARY OUTCOMES:
Barthel's index | On day 1, and at 90 days
  An improvement of 10 or more points in Barthel's index will be considered a favorable outcome.
NIH stroke scale score | On day 1, day 4 or discharge whichever is earlier, and at 90 days
Depression score using the PHQ9 questionnaire | On day 1, and day 4 or discharge whichever is earlier.
Infarct volumes | On day 1, and day 4 or discharge whichever is earlier
  Measured from the DWI-MRI and/or CT images
All cause mortality | 90 days
Stroke-related mortality | 90 days
Symptomatic intracranial hemorrhage | Day 4 or discharge whichever is earlier
Deterioration in neurologic status | Up to day 4 or discharge whichever is earlier
  Increase of 4 or more points in the NIH stroke scale

CONTACTS AND LOCATIONS:
Locations (1):
- Lankenau Medical Center, Wynnewood, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No